CLINICAL TRIAL: NCT00367445
Title: A 1 Month, Open-Label Inpatient, Randomized Cross-Over Trial Assessing The Impact Of Dry Powder Inhaled Insulin (Exubera) On 24-Hour Glycemic Control Compared To Insulin Glargine (Lantus) In Patients With Type 2 Diabetes Mellitus Who Are Poorly Controlled On A Combination Of Two Oral Agents
Brief Title: A Clinical Trial Comparing Short-Term Efficacy and Safety of Exubera and Lantus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A2171094
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exubera; Insulin Glargine

INTERVENTIONS:
Drug: Inhaled Human Insulin (Exubera)
Drug: Insulin Glargine (Lantus)

SUMMARY:
To compare short-term efficacy and safety of Exubera vs Lantus in patients with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus Type 2

Exclusion Criteria:

* Severe Asthma, severe COPD
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-09; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Variability of blood glucose over a period of 72 hours

SECONDARY OUTCOMES:
Insulin pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Chula Vista, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171094&StudyName=A+Clinical+Trial+Comparing+Short%2Dterm+Efficacy+and+Safety+of+Exubera+and+Lantus